CLINICAL TRIAL: NCT03650504
Title: Effects of Catheter Location Relative to Femoral Artery on Postoperative Analgesia for Continuous Adductor Canal Blocks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: Rodney Gabriel MD (Unknown); Matthew Swisher MD (Unknown)
Responsible Party: Principal Investigator, John J. Finneran IV, MD, Assistant Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 180718
Record Dates: First submitted 2018-08-22; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Above Artery Group (Experimental)
  Interventions: Procedure: Above Artery Catheter Placement
- Between Artery and Vein Group (Active Comparator)
  Interventions: Procedure: Between Artery and Vein Placement

INTERVENTIONS:
Procedure: Above Artery Catheter Placement — Nerve catheter placed between superficial femoral artery and sartorial muscle
  Arms: Above Artery Group
Procedure: Between Artery and Vein Placement — Nerve catheter placed between superficial femoral artery and femoral vein
  Arms: Between Artery and Vein Group

SUMMARY:
Adductor canal (AC) nerve block is a commonly used modality for postoperative pain control after total knee arthroplasty (TKA). When the adductor canal is viewed by ultrasound, the femoral artery and femoral vein can easily be identified, however, the nerve that is to be blocked is often not visible. For this reason, the femoral artery is used as a landmark for the block. There currently are no studies examining the optimal placement of the nerve block catheter relative to the femoral artery in the canal. The goal of this study will be to examine the relationship between nerve catheter tip location relative to femoral artery within the adductor canal for continuous AC nerve blocks. The investigators specifically will compare postoperative pain as well as incidence of vascular puncture during the procedure and time to complete the procedure for two different catheter locations.

DETAILED DESCRIPTION:
This will be a single-center, randomized, controlled investigation. Consenting adults undergoing unilateral total knee arthroplasty with a planned adductor canal perineural catheter will be offered enrollment. Study inclusion will be proposed to eligible patients prior to surgery. If a patient desires study participation, written, informed consent will be obtained using a current UCSD IRB-approved ICF. Selection for inclusion will not be based on gender, race, or socioeconomic status.

Following written, informed consent, we will record baseline anthropomorphic information. All subjects will have a peripheral intravenous (IV) catheter inserted, standard noninvasive monitors applied, supplemental oxygen administered via a nasal cannula or face mask, and positioned supine. Midazolam and fentanyl will be titrated for patient comfort, while ensuring that patients remain responsive to verbal cues. The ultrasound will be placed to visualize the short axis (cross-section) of the adductor canal. If both sites (above femoral artery versus between femoral artery and vein) are acceptable for catheter insertion, the subject will be randomized using a computer-generated list (blocks of 8) to one of two treatment groups in a 1:1 ratio using sealed, opaque, consecutively numbered envelopes: (1) above femoral artery vs (2) between femoral artery and vein.

Catheter insertion will adhere to current UCSD standard-of-care. The only difference for subjects participating in the study will be that the specific catheter insertion location will be determined randomly, instead of the physician simply choosing him/herself. All catheters will be placed by a regional anesthesia fellow under the direct supervision and guidance of a regional anesthesia attending. All catheters will be placed using standard UCSD perineural catheter techniques.

The area of insertion will be cleaned with chlorhexidine gluconate and isopropyl alcohol, and a clear, sterile, fenestrated drape applied. The ultrasound probe will be placed to visualize the short-axis (cross-section) of the target nerve(s). A 17-gauge needle (FlexTip, Teleflex Medical, Triangle Research Park, NC, USA) will be used to place all perineural catheters. The catheter-placement needle will be inserted through the skin wheal, advanced in-plane beneath the US transducer and directed to the target nerve as described below:

"Above-the-artery": The needle will be directed below the nerve to about five o'clock of the artery. The needle will then be advanced to twelve o'clock of the artery while opening the adductor canal space with saline until adequate opening of the canal is realized. At that point, the catheter is placed above the artery.

"Between-the-artery-and-vein": The needle will be directed above the nerve and placed at one o'clock of the artery. Then the needle will be positioned at about six o'clock of the artery and advanced between the femoral artery and vein with simultaneous pressure until the adductor canal opens appropriately. The perineural catheter will be placed between the artery and vein.

Saline (10 mL) will be administered via the needle to dilate the space where the catheter is to be inserted. A flexible non-stimulating perineural catheter will be inserted 3-5 cm past the needle tip; and the needle withdrawn over the catheter. A 30 mL bolus of lidocaine 2% with 1:400,000 of epinephrine will then be administered through the catheter.

Intraoperatively, patients may receive a general and/or neuraxial anesthetic that would be determined by the intraoperative anesthesia provider. Additional boluses of 10 mL 2% lidocaine with epinephrine may be given, if needed, via the perineural catheter.

Perineural infusion: An infusion pump will be attached to each subject's perineural catheter. The pump will provide ropivacaine 0.2% at 6 mL/h and a 4 mL patient-controlled bolus with a 30-minute lockout.

Data collection: All data collection will be through standard UCSD nursing/therapy electronic medical record notes for the day following surgery.

Primary endpoint: The primary endpoint will be the average pain on post operative day 1 following surgery as measured on a numeric rating scale (0-10, 0=no pain, 10=worst imaginable pain) during the time periods of 08:00-24:00.

Secondary endpoints: Other data collected will include: (1) total procedure duration (from needle-in to needle-out), (2) total opioid consumption on postoperative day 1, (3) worst pain score measured on a numeric rating scale, (4) number of intra-procedural vascular punctures, (5) total local anesthetic infused in 24 hours following surgery, and (6) distance ambulated on postoperative day 1 with first session of physical therapy.

Sample size estimates:

The primary analysis will utilize the Wilcoxon Rank Sum test. The mean postoperative day 1 pain scores following adductor canal catheter placement for total knee arthroplasty is 4.12 with standard deviation = 1.74.2 The null hypothesis is that the "above-the-artery" group is inferior to the "between-the-artery-and-vein" group. The alternative hypothesis is that the "above-the-artery" group in non-inferior to the "between-the-artery-and-vein" group. Assuming a non-inferiority limit of 1.5, power = 0.80, two-side alpha = 0.05, we will require 17 patients in each group (total = 34). To account for dropouts, we plan to recruit 20 patients in each group, totaling 40 patients all together.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral total knee arthroplasty at UC San Diego with planned placement of an adductor canal catheter at request of surgeon

Exclusion Criteria:

* history of allergic reaction to lidocaine or ropivacaine
* history of peripheral neuropathy, neuropathic pain, or chronic pain requiring opioid medications.
* Pregnant females and prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-24 (Estimated); Primary Completion 2019-07-30 (Estimated); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
AVERAGE PAIN | 08:00AM to 24:00 on the first day following surgery
  Average pain on post operative day 1 following surgery as measured on a numeric rating scale (0-10, 0=no pain, 10=worst imaginable pain).

SECONDARY OUTCOMES:
Procedure duration | Prior to surgery
Opioid consumption | Postoperative days zero and one
Distance Ambulated | Physical Therapy sessions on postoperative day one
Worst pain score (NRS 0-10 reported by patient) | Postoperative day , entire day
Number of vascular pictures during placement | During the catheter placement procedure
Intravascular injection assessed by heart rate response to epinephrine in injection | During the catheter placement procedure
Total local anesthetic infused on first postoperative day | Postoperative days zero and one

IPD SHARING:
Plan to Share IPD: No